CLINICAL TRIAL: NCT00003595
Title: Randomized Trial of CHOP Chemotherapy With or Without Rituximab (Chimeric Anti-CD20 Antibody) for HIV-Associated Non-Hodgkin's Lymphoma
Brief Title: Combination Chemotherapy With or Without Monoclonal Antibody Therapy in Treating Patients With Previously Untreated HIV-Associated Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02279; AMC-010; CPMC-IRB-9691; CWRU-AMC-1400; UCLA-9810029; CDR0000066666 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2003-10-28 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2007-05

CONDITIONS: Lymphoma
Keywords: childhood Burkitt lymphoma; AIDS-related peripheral/systemic lymphoma; AIDS-related diffuse large cell lymphoma; AIDS-related immunoblastic large cell lymphoma; AIDS-related small noncleaved cell lymphoma
MeSH Terms: conditions — Lymphoma; Burkitt Lymphoma | interventions — Filgrastim; Rituximab; VAP-cyclo protocol; Cyclophosphamide; Doxorubicin; Prednisone; Vincristine

ARMS (2):
- Arm I (Experimental): Patients receive cyclophosphamide IV, doxorubicin IV, and vincristine IV on day 3 and oral prednisone on days 3-7. Patients receive rituximab on day 1. Treatment repeats every 3 weeks for a minimum of 4 courses or 2 courses beyond complete response in the absence of disease progression or unacceptable toxicity. Patients with stage I, stage IE (including bulky), or nonbulky stage II or IIE disease receive 3 courses of chemotherapy with rituximab followed by radiotherapy beginning 3 weeks after completion of the third course. Patients who achieve partial response for a minimum of 28 days or complete response receive maintenance rituximab IV beginning on day 28 of the final course of chemotherapy. Maintenance rituximab treatment repeats every 4 weeks for 3 courses.
  Interventions: Biological: filgrastim; Biological: rituximab; Drug: CHOP regimen; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: prednisone; Drug: vincristine sulfate
- Arm II (Active Comparator): Patients receive cyclophosphamide IV, doxorubicin IV, and vincristine IV on day 1 and oral prednisone on days 1-5. Treatment repeats every 3 weeks for a minimum of 4 courses or 2 courses beyond complete response. Patients with stage I, stage IE (including bulky), or nonbulky stage II or IIE disease receive 3 courses of chemotherapy. Patients receive radiotherapy beginning 3 weeks after completion of the third course of chemotherapy.
  Interventions: Biological: filgrastim; Drug: CHOP regimen; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: prednisone; Drug: vincristine sulfate

INTERVENTIONS:
Biological: filgrastim
Biological: rituximab
  Arms: Arm I
Drug: CHOP regimen
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: prednisone
Drug: vincristine sulfate

SUMMARY:
Randomized phase III trial to compare the effectiveness of combination chemotherapy with or without monoclonal antibody therapy in treating patients who have previously untreated HIV-associated non-Hodgkin's lymphoma. Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Monoclonal antibodies such as rituximab can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. It is not yet known whether combination chemotherapy plus monoclonal antibody therapy is more effective than combination chemotherapy alone in treating HIV-associated non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Compare the efficacy of CHOP (cyclophosphamide, doxorubicin, vincristine, and prednisone) with or without rituximab in patients with previously untreated HIV-associated non-Hodgkin's lymphoma.

II. Determine the efficacy of rituximab as maintenance therapy following remission induction with CHOP in these patients.

III. Determine the effect of rituximab on the immune system and HIV viral load in these patients.

IV. Determine the relationship between EBV load and the presence of EBV in lymphoma tumor cells of these patients.

V. Compare the effect of CHOP with or without rituximab on EBV load in these patients.

OUTLINE: This is a randomized, multicenter study.

Patients are stratified by extent of disease (stage I/II vs III/IV). Patients are randomized to 1 of 2 treatment arms:

Arm I: Patients receive cyclophosphamide IV, doxorubicin IV, and vincristine IV on day 3 and oral prednisone on days 3-7. Patients receive rituximab on day 1. Treatment repeats every 3 weeks for a minimum of 4 courses or 2 courses beyond complete response in the absence of disease progression or unacceptable toxicity. Patients with stage I, stage IE (including bulky), or nonbulky stage II or IIE disease receive 3 courses of chemotherapy with rituximab followed by radiotherapy beginning 3 weeks after completion of the third course. Patients who achieve partial response for a minimum of 28 days or complete response receive maintenance rituximab IV beginning on day 28 of the final course of chemotherapy. Maintenance rituximab treatment repeats every 4 weeks for 3 courses.

Arm II: Patients receive cyclophosphamide IV, doxorubicin IV, and vincristine IV on day 1 and oral prednisone on days 1-5. Treatment repeats every 3 weeks for a minimum of 4 courses or 2 courses beyond complete response. Patients with stage I, stage IE (including bulky), or nonbulky stage II or IIE disease receive 3 courses of chemotherapy. Patients receive radiotherapy beginning 3 weeks after completion of the third course of chemotherapy.

Both arms: Patients receive filgrastim (G-CSF) subcutaneously beginning on day 4 and continuing through day 13 of each chemotherapy course or until blood counts recover.

Patients are followed every 4 weeks for 1 year and then every 2 months until death.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically proven HIV-associated B cell non-Hodgkin's lymphoma, including:
* Diffuse large B cell lymphoma
* Intermediate grade diffuse large cell lymphoma
* High grade large cell immunoblastic lymphoma
* Burkitt's lymphoma
* High grade B cell lymphoma, Burkitt's like (small noncleaved lymphoma)
* No primary CNS lymphoma (parenchymal brain or spinal cord tumor)
* Evaluable disease HIV documentation may be serologic (ELISA or western blot), culture, or quantitative PCR or bDNA assay Tumors must be CD20 positive (greater than 50% cells express CD20)
* A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS:

* Age: Over 18
* Performance status: Karnofsky 70-100%
* Absolute neutrophil count greater than 1,000/mm3*
* Platelet count greater than 75,000/mm3*

  * Unless cytopenias are secondary to lymphoma
* Bilirubin less than 2.0 mg/dL (unless secondary to hepatic infiltration with lymphoma or isolated hyperbilirubinemia associated with the use of indinavir)
* SGOT or SGPT less than 7 times upper limit of normal
* Creatinine less than 2.0 mg/dL (unless due to lymphoma)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No acute, active HIV-associated opportunistic infection requiring antibiotics
* Mycobacterium avium complex allowed
* No concurrent malignancy except carcinoma in situ of the cervix, nonmetastatic nonmelanomatous skin cancer, or Kaposi's sarcoma not requiring systemic chemotherapy

PRIOR CONCURRENT THERAPY:

* Prior or concurrent epoetin alfa or filgrastim (G-CSF) allowed
* No prior colony stimulating factor therapy within 24 hours prior to chemotherapy
* No prior chemotherapy for HIV-associated non-Hodgkin's lymphoma
* At least 1 year since prior cyclophosphamide or doxorubicin
* No prior radiotherapy for HIV-associated non-Hodgkin's lymphoma
* Chronic therapy with myelosuppressive agents allowed
* Concurrent antiretroviral therapy, antifungal medications, and antibiotics allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 1999-01; Primary Completion 2006-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence D. Kaplan, MD, Study Chair — University of California, San Francisco
Locations (13):
- United States (13):
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - San Francisco General Hospital Medical Center, San Francisco, California
  - Sylvester Cancer Center, University of Miami, Miami, Florida
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - University Hospital/New Jersey Cancer Center, Newark, New Jersey
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Ireland Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio

REFERENCES:
- [Background] Chadburn A, Chen X, Chiu A, et al.: Neither germinal center (GC) vs non-germinal center (Non-GC) phenotype nor FOXP1 expression correlate with outcome in AIDS-associated diffuse large B-cell lymphoma (DLBCL): study of patients from AIDS Malignancies Consortium trials 010 and 034. [Abstract] Blood 108 (11): A-2023, 2006.
- [Result] Chen X, Cesarman E, Hyjek E, et al.: FOXP1 expression in AIDS-associated diffuse large B-cell lymphoma (DLBCL): correlation with prognostic parameters in patients from AIDS Malignancies Consortium Trial 010. [Abstract] United States and Canadian Academy of Pathology 95th Annual Meeting, February 11-17, 2006, Atlanta, GA. A-1016, 2006.
- [Result] Kaplan LD, Lee JY, Ambinder RF, Sparano JA, Cesarman E, Chadburn A, Levine AM, Scadden DT. Rituximab does not improve clinical outcome in a randomized phase 3 trial of CHOP with or without rituximab in patients with HIV-associated non-Hodgkin lymphoma: AIDS-Malignancies Consortium Trial 010. Blood. 2005 Sep 1;106(5):1538-43. doi: 10.1182/blood-2005-04-1437. Epub 2005 May 24. PMID 15914552